CLINICAL TRIAL: NCT02884414
Title: Analysis of Joint Mechanics in Response to Gait Modifications and Cutaneous Stimulation
Brief Title: Gait Modifications and Cutaneous Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Peter Andriacchi, Principal Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 37562
Record Dates: First submitted 2016-08-23; First posted 2016-08-31 (Estimated); Results first posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee Pathology
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cutaneous Stimulation (Experimental): Cutaneous stimulation and/or feedback. This stimulation and/or feedback may be visual, auditory, tactile (e.g. vibratory, temperature), or haptic and is completely external.
  Interventions: Device: Cutaneous stimulation

INTERVENTIONS:
Device: Cutaneous stimulation — A non-invasive external device that will be placed on the leg of the subject. The device consists of a sensing module to determine specific points in the gait cycle, a processor to analyze signal from the sensor, and a stimulus module to provide feedback to the subject.

SUMMARY:
The purpose of this study is to quantify differences in joint mechanics between different types of walking in healthy individuals and individuals with knee pathology. The investigators will determine how modifying gait through feedback and/or cutaneous stimulation changes joint loading.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 35 kg/m^2
* For knee pathology subjects: Diagnosis of knee pathology (e.g. knee osteoarthritis, ACL injury, etc) and/or knee pain
* Full weight-bearing status

Exclusion Criteria:

* Non-ambulatory
* Use of walking aid
* For healthy volunteers - history of surgical intervention at any joint of the lower extremity
* Inability to cooperate with study protocol due to medical or psychiatric reasons
* Inability to provide informed consent
* For healthy subjects: Any diagnosis of knee osteoarthritis or knee pain

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-08; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Andriacchi, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cutaneous Stimulation
Started | 56
Completed | 56
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cutaneous Stimulation
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (18.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 17
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 36
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 56
Knee Flexion Moment [Mean (Standard Deviation); unit: %Bw*Ht] — The peak knee flexion moment during stance phase of gait, collected during motion capture analysis at a self-selected normal walking speed. Population: Data excluded from n=3 participants due to technical data collection issue.
  %Bw*Ht
    number analyzed (Participants) | 53
    (all) | 2.68 (1.29)

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak Knee Flexion Moment (%Bw*Ht)
Description: Within-subject change in peak knee flexion moment (%Bodyweight*Height) with the intervention versus control (without the intervention).
Time Frame: Immediate
Measure: Mean (Standard Deviation); unit: %Bw*Ht
Arm/Group | Cutaneous Stimulation
Number analyzed (Participants) | 53
%Bw*Ht | 2.72 (1.25)
Statistical Analysis 1: Comparison: Cutaneous Stimulation; Test type: Other — Paired Student's t-test; p = 0.44, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: During the day of study participation.
Arm/Group | Cutaneous Stimulation
All-Cause Mortality (participants affected / at risk) | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56
Other Adverse Events (participants affected / at risk) | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-02): https://cdn.clinicaltrials.gov/large-docs/14/NCT02884414/Prot_SAP_000.pdf